CLINICAL TRIAL: NCT05155176
Title: Novel Methods for Investigating Stress-related Processes in Social Drinkers and Individuals With Alcohol Use Disorder
Brief Title: Novel Real-world Methods in Social Drinkers and AUD
Acronym: ALR
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Peter McManus Charitable Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2000031842
Record Dates: First submitted 2021-12-07; First posted 2021-12-13 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Alcohol Drinking; Alcohol Abuse; Alcohol Use Disorder
Keywords: Alcohol Use Disorder; Smartphone; Alcohol; Cortisol; Heart rate variability; Ecological Momentary Assessment
MeSH Terms: conditions — Alcohol Drinking; Alcoholism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with Alcohol Use Disorder: Participants who meet the criteria for Alcohol Use Disorder will complete six weeks of smartphone monitoring. During this monitoring period, they will also complete two three-consecutive days of intensive monitoring including more frequent smartphone surveys, saliva samples, heart rate monitoring, and an alcohol use monitor.
  Interventions: Behavioral: Intensive Day Monitoring
- Social drinkers: Participants who have a past year history of alcohol use and do not meet the criteria for Alcohol Use Disorder will complete two weeks of smartphone monitoring. During this monitoring period, they will also complete three consecutive days of intensive monitoring including more frequent smartphone surveys, saliva samples, heart rate monitoring, and an alcohol use monitor.
  Interventions: Behavioral: Intensive Day Monitoring

INTERVENTIONS:
Behavioral: Intensive Day Monitoring — During intake, a research assistant will demonstrate how to place the HRV monitor, BACtrak Skyn, and provide instructions on completing the saliva samples at home. Participants will wear the HRV and Skyn monitors for three consecutive, randomly selected days twice for individuals with Alcohol Use Disorder and once for social drinkers during the study (72 hours each). Participants will be provided with six saliva sample collection tubes per day with explicit directions on when the saliva sampling should occur (hours since waking: +0, +1, +2, +4, +6, +10 hours, and before going to sleep). Participants will also complete a subjective report using similar questions included in the survey prompts at the same scheduled time as the saliva sample. Individuals with Alcohol Use Disorder would complete a total of 6 such days during the study, and social drinkers would complete a total of 3 such days during the study.

SUMMARY:
This research project proposes a novel approach to elucidate the biological adaptations associated with Alcohol Use Disorder and to assess whether such adaptations are predictive of higher alcohol craving in response to both alcohol cues and stressors and higher relapse risk and alcohol use in the real world.

DETAILED DESCRIPTION:
We will use intensive longitudinal data collection and analysis across multiple data streams. We will recruit 25 treatment-seeking individuals with AUD and 25 light social drinkers matched on demographically relevant variables (i.e., age, gender, IQ, race). We will use smartphones to assess subjects' alcohol use and experiences in real-time via ecological momentary assessment (EMA). During three consecutive days of these two weeks, we propose using passive biomonitoring to collect real-time cardiovascular responses, i.e., heart rate variability (HRV), and alcohol use via unobtrusive monitors (i.e., Firstbeat Bodyguard 2, BACtrack Skyn) with scheduled salivary cortisol samples. Individuals with AUD will then be provided with four weeks of behavioral treatment with daily assessments. During the final two weeks of treatment, individuals with AUD will complete another three-day period of intensive self-reports, including another 72-hours physiological and salivary cortisol monitoring.

ELIGIBILITY:
Inclusion Criteria:

Men and women who:

1) Are older than 18 years old at the first intake appointment; 2) Are fluent in English; 3) Are drinking alcohol at levels to match either of the two groups:

a. Social drinkers: i. Must report a past-year history of alcohol use ii. Must not meet current AUD and may have only met mild AUD during their lifetime (not within the past year) iii. Provide a negative urine toxicology screen. b. Individuals with Alcohol Use Disorder: i. Must meet current criteria for AUD based on the SCID (≤ 2 symptoms in past year); ii. Report at least weekly use of alcohol. iii. Do not meet criteria for any other substance use disorders other than mild Cannabis Use Disorder.

iv. Provide a positive urine toxicology screen for alcohol during intake. 5) Can provide written informed consent.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1. Meets current or past DSM-5 criteria for Axis I for major psychiatric disorders, other than depression or anxiety disorder;
  2. Meets criteria for a current Substance Use Disorder other than Alcohol or mild Cannabis Use Disorder;
  3. Has any significant current medical conditions requiring medication, including neurological, renal, thyroid, cardiovascular, liver, endocrine, or immune conditions;
  4. Reports current use of medications/drugs that interfere with HPA axis response,
  5. Are women who are pregnant or lactating;
  6. Report current use of psychotropic drugs other than antidepressants.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Rating of subjective craving in the real world | 42 days for individuals with AUD, 14 days for social drinkers
  Participants will report using ecological momentary assessment (EMA) their current levels of craving, if they have drank alcohol, and if they experienced a stressor. These reports will be generated in three different ways: at 8 am and 8 pm at night, at four random times during waking hours, and while drinking alcohol. Individuals with AUD will be compared to social drinkers in their differences in real-world ratings of stress and craving. Craving and stress will be assessed using a 100-point visual analog scale (VAS) in which 0="Not at all" and 100="Extremely High."
Rating of subjective stress in the real world | 42 days for individuals with AUD, 14 days for social drinkers
  Participants will report using ecological momentary assessment (EMA) their current levels of stress, if they have drank alcohol, and if they experienced a stressor. These reports will be generated in three different ways: at 8 am and 8 pm at night, at four random times during waking hours, and during marijuana use. Individuals with AUD will be compared to social drinkers in their differences in real-world ratings of stress and craving. Craving and stress will be assessed using a 100-point visual analog scale (VAS) in which 0="Not at all" and 100="Extremely High."
Heart rate response to stress and cannabis cues in the real world | 6 days for individuals with AUD, 3 days for social drinkers
  Heart Rate Variability (HRV) will be collected throughout the day on two (individuals with AUD) or one set (social drinkers) of three-day occasions during intake week and during week 6 of the study.
Cortisol response to stress and cannabis cues in the real world | 6 days for individuals with AUD, 3 days for social drinkers
  Saliva samples for cortisol levels will be collected throughout the day on two (individuals with AUD) or one set (social drinkers) of three-day occasions during intake week and during week 6 of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Wemm, PhD, Principal Investigator — Yale University
Locations (1):
- Yale Stress Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No